CLINICAL TRIAL: NCT03683537
Title: Association Between Changes of GFAP After Surgery and Postoperative Delayed Cognitive Recovery
Status: Completed | Type: Observational
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Other Study IDs: MKNC 02/2018
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Astrogliosis; Postoperative Cognitive Dysfunction; Postoperative Delirium
MeSH Terms: conditions — Gliosis; Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Delayed Neurocognitive decline: Patients in whom there is Delayed Neurocognitive Recovery (DNR) after surgery, based on neuropsychological tests or clinically. DNR is defined as follow: 1)decrease of scores of neuropsychological test scores for more than 1 standard deviation (SD) of these tests; 2)clinically - inability of patient to perform test after surgery because of neurocognitive impairment.
  Interventions: Diagnostic Test: Glial fibrillary acidic protein
- Normal postop neurocognitive function: Patients in whom there is no clinical signs of DNR, defined as in previous group.
  Interventions: Diagnostic Test: Glial fibrillary acidic protein

INTERVENTIONS:
Diagnostic Test: Glial fibrillary acidic protein — 3 samples of serum are drawn from patients. The 1st Sample of patient serum is drawn before induction into anesthesia. The 2nd is drawn 24 hours after the 1st one. The 3rd sample is drawn on 3 or 4 postoperative day. All samples collected and preserved in the same temperature as required for ELISA.

SUMMARY:
Assessment of serum level of glial fibrillary acidic protein (GFAP) before surgery (on the day of surgery), 24 hours after surgery and on 3 or 4 postoperative day. Neuropsychological testing before surgery and on 3 or 4 day after surgery. Investigation of relationship between changes of GFAP and scores of neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with different diseases, who require prolonged laparoscopy or open surgery
* Age more than 60
* ASA I-III
* Informed consent to participate in the study

Exclusion Criteria:

* ASA IV-V
* Severe neurodegenerative or psychological diseases

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo surgery in Moscow Clinical Scientific Center
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in serum GFAP | 1 year
  GFAP(3) - GFAP (1); GFAP (2) - GFAP (1)

CONTACTS AND LOCATIONS:
Overall Officials: Valery Subbotin, Ph.D., M.D., Study Chair — Moscow Clinical Scintific Center
Locations (1):
- Moscow Clinical Scientific Center, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided